CLINICAL TRIAL: NCT04266028
Title: A Randomized, Double-blind, Placebo-controlled, Dose Escalation Study to Evaluate the Safety and Tolerability of Subcutaneous Immunotherapy With DM-101 in Adults With Birch Pollen Allergy
Brief Title: Study to Evaluate Safety and Tolerability of sc Immunotherapy With DM-101 in Adults With Birch Pollen Allergy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Desentum Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: DM-101-C-001; 2019-001936-67 (EudraCT Number)
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2021-06

CONDITIONS: Birch Pollen Allergy

STUDY DESIGN:
Intervention Model Description: 4 sequential study cohorts with ascending DM-101 doses. In each cohort two treatment arms: placebo and active drug
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- DM-101 Single Dose (Experimental): Participants received a single subcutaneous (SC) dose of DM-101 30 ng on Day 1
  Interventions: Biological: DM-101
- Placebo Single Dose (Placebo Comparator): Participants received a single SC injection of placebo on Day 1
  Interventions: Biological: Placebo to match DM-101
- DM-101 Low Multiple Ascending Doses (MAD) (Experimental): Participants received 5 biweekly administered SC doses of DM-101 as follows: 30 ng on Day 1,50 ng on Day 14, 100 ng on Day 28, 42, and 56.
  Interventions: Biological: DM-101
- Placebo Low MAD (Placebo Comparator): Participants received 5 biweekly administered SC injections of placebo on Day 1,14, 28, 42, and 56.
  Interventions: Biological: Placebo to match DM-101
- DM-101 High MAD (Experimental): Participants received 5 biweekly administered SC doses of DM-101 as follows: 30 ng on Day 1,50 ng on Day 14, 100 ng on Day 28, 200 ng (dose divided into two SC injections) on Day 42, and 300 ng (dose divided into three SC injections) on Day 56.
  Interventions: Biological: DM-101
- Placebo High MAD (Placebo Comparator): Participants received 5 biweekly administered SC injections of placebo as follows: single injection on Day 1, 14 and 28; two injections on Day 42; three injections on Day 56.
  Interventions: Biological: Placebo to match DM-101
- DM-101 2-Day Ultra-Rush Dose Escalation (Experimental): Participants received 9 SC doses of DM-101 as follows: 100, 250, 500, 1000, 2500, 5000, 10000 and 25000 ng during Day 1 and Day 2.
  Interventions: Biological: DM-101
- Placebo 2-Day Ultra-Rush Dose Escalation (Placebo Comparator): Participants received 9 SC injections of placebo during Day 1 and Day 2.
  Interventions: Biological: Placebo to match DM-101

INTERVENTIONS:
Biological: DM-101 — DM-101 administered by subcutaneous (SC) injection
  Arms: DM-101 2-Day Ultra-Rush Dose Escalation; DM-101 High MAD; DM-101 Low Multiple Ascending Doses (MAD); DM-101 Single Dose
Biological: Placebo to match DM-101 — Placebo to match DM-101 administered by SC injection
  Arms: Placebo 2-Day Ultra-Rush Dose Escalation; Placebo High MAD; Placebo Low MAD; Placebo Single Dose

SUMMARY:
Randomized, double-blind placebo-controlled phase I study to investigate the safety and tolerability of ascending doses of DM-101 in adult subjects with birch pollen allergy.

DETAILED DESCRIPTION:
The study will be carried out in a single study site located in Finland.

ELIGIBILITY:
Key Inclusion Criteria:

* Males or females, aged 18 to 65 years
* Good general health
* A documented clinical history of birch pollen-induced allergic rhinitis or rhinoconjunctivitis with symptoms that interfere with daily activities or sleep and remain bothersome despite the use of relevant symptomatic medication, and have been present over, at least, 2 allergy seasons.
* Bet v 1 specific serum IgE ≥ 0.7 kU/L
* Positive SPT to birch pollen allergen, with a wheal diameter ≥ 5 mm
* Body weight ≥50 kg and body mass index (BMI) within the range 18-35 kg/m2.

Key Exclusion Criteria:

* History or findings on physical examination of any significant disease or disorder which, in the opinion of the Investigator, may put the subject at risk because of participation in the study, influence the results of the study or the subject's ability to participate in the study.
* Current diagnosis of asthma (other than seasonal during the birch pollen allergy season), requiring Global Initiative for Asthma (GINA) Step 2 or higher treatment, or asthma partially controlled or uncontrolled according to GINA classification in the 6 months before Screening.
* History of asthma deterioration that resulted in emergency treatment or hospitalisation in the 12 months before screening, or a life-threatening asthma attack at any time in the past.
* Forced Expiratory Volume in one second (FEV1) < 70% of predicted, regardless of asthma status at screening or baseline assessment at the first dosing visit.
* History of severe drug allergy, severe angioedema or systemic allergic reaction of Grade 3 or greater, according to the World Allergy Organization (WAO) scale, due to any cause.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Nilson, Study Director — Desentum Oy; Mika Scheinin, Principal Investigator — Clinical Research Services Turku
Locations (1):
- Clinical Research Services Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to patient level data and related study documents. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants after Desentum has received marketing authorization from major health authorities (e.g., FDA, EMA), has the legal authority to share the data, and has made the study results publicly available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at one study site in Finland. The first participant was screened 11 February 2020. The last study visit occurred on 31 Mat 2021.
Pre-assignment Details: 61 participants were screened.
Period: Overall Study
Arm/Group | DM-101 Single Dose | Placebo Single Dose | DM-101 Low Multiple Ascending Doses (MAD) | Placebo Low MAD | DM-101 High MAD | Placebo High MAD | DM-101 2-Day Ultra-Rush Dose Escalation | Placebo 2-Day Ultra-Rush Dose Escalation
Started | 4 | 2 | 6 | 2 | 6 | 2 | 4 | 1
Completed | 4 | 2 | 5 | 2 | 4 | 2 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 2 | 0 | 4 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Not completed — temporary halt of the study | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Onset of birch pollen season | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | DM-101 Single Dose | Placebo Single Dose | DM-101 Low Multiple Ascending Doses (MAD) | Placebo Low MAD | DM-101 High MAD | Placebo High MAD | DM-101 2-Day Ultra-Rush Dose Escalation | Placebo 2-Day Ultra-Rush Dose Escalation | Total
Number analyzed (Participants) | 4 | 2 | 6 | 2 | 6 | 2 | 4 | 1 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (10.81) | 27.5 (4.95) | 29.8 (11.34) | 26.5 (4.95) | 37.7 (8.43) | 34.5 (7.78) | 44.0 (5.03) | 33.0 (0.0) | 31.11 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 5 | 2 | 2 | 1 | 2 | 1 | 15
  Male | 2 | 2 | 1 | 0 | 4 | 1 | 2 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6 | 2 | 6 | 2 | 4 | 1 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 2 | 6 | 2 | 6 | 2 | 4 | 1 | 27
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Finland | 4 | 2 | 6 | 2 | 6 | 2 | 4 | 1 | 27

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events
Description: Number of All Treatment Emergent Adverse Events (TEAEs) in Subjects Receiving DM-101 Compared to Placebo
Time Frame: From the first dose until 28 days following the last dose.
Population: The Safety Set included participants who received at least 1 dose of study drug.
Measure: Number; unit: number of adverse events per arm
Arm/Group | DM-101 Single Dose | Placebo Single Dose | DM-101 Low Multiple Ascending Doses (MAD) | Placebo Low MAD | DM-101 High MAD | Placebo High MAD | DM-101 2-Day Ultra-Rush Dose Escalation | Placebo 2-Day Ultra-Rush Dose Escalation
Number analyzed (Participants) | 4 | 2 | 6 | 2 | 6 | 2 | 4 | 1
number of adverse events per arm | 13 | 3 | 81 | 2 | 88 | 7 | 72 | 2
Statistical Analysis 1: Comparison: DM-101 Single Dose vs Placebo Single Dose vs DM-101 Low Multiple Ascending Doses (MAD) vs Placebo Low MAD vs DM-101 High MAD vs Placebo High MAD vs DM-101 2-Day Ultra-Rush Dose Escalation vs Placebo 2-Day Ultra-Rush Dose Escalation; No statistical analyses were performed; Test type: Other — No statistical analyses were performed; No statistical analyses were performed; no statistical analyses were performed = 0; No statistical analyses were performed

2. Secondary Outcome: Number and Severity of Systemic Allergic Reactions (SARs) in Subjects Receiving DM-101 Compared to Placebo
Description: Severity of SARs are graded from Grade 1 to 5 (Grade 5 being fatal) as defined by WAO Subcutaneous Immunotherapy Systemic Reaction Grading System.
Time Frame: From the first dose until 28 days following the last dose.
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Number; unit: number of systemic reactions per arm
Arm/Group | DM-101 Single Dose | Placebo Single Dose | DM-101 Low Multiple Ascending Doses (MAD) | Placebo Low MAD | DM-101 High MAD | Placebo High MAD | DM-101 2-Day Ultra-Rush Dose Escalation | Placebo 2-Day Ultra-Rush Dose Escalation
Number analyzed (Participants) | 4 | 2 | 6 | 2 | 6 | 2 | 4 | 1
number of systemic reactions per arm
  Grade 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number and Severity of Local Injection Site Reactions (LISRs) in Subjects Receiving DM-101 Compared to Placebo
Description: Pain, tenderness, erythema/redness and induration/swelling at the injection site was assessed after each injection using a 4-point scale (Grade 1 = mild, Grade 4 = severe) as defined in the study protocol.
Time Frame: From the first dose until 28 days following the last dose.
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: number of LISRs per arm
Arm/Group | DM-101 Single Dose | Placebo Single Dose | DM-101 Low Multiple Ascending Doses (MAD) | Placebo Low MAD | DM-101 High MAD | Placebo High MAD | DM-101 2-Day Ultra-Rush Dose Escalation | Placebo 2-Day Ultra-Rush Dose Escalation
Number analyzed (Participants) | 4 | 2 | 6 | 2 | 6 | 2 | 4 | 1
number of LISRs per arm
  Grade 1 | 4 | 0 | 26 | 1 | 27 | 0 | 3 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 8 | 0 | 12 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Subjects Reaching the Pre-defined DM-101 Dose
Description: Proportion of subjects reaching the pre-defined, admissible dose in each DM-101 dosing group
Time Frame: From the first dose until 28 days following the last dose.
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | DM-101 Single Dose | DM-101 Low Multiple Ascending Doses (MAD) | DM-101 High MAD | DM-101 2-Day Ultra-Rush Dose Escalation
Number analyzed (Participants) | 4 | 6 | 6 | 4
Participants | 4 | 5 | 4 | 0

ADVERSE EVENTS:
Time Frame: From the first dose until 28 days following the last dose
Arm/Group | DM-101 Single Dose | Placebo Single Dose | DM-101 Low Multiple Ascending Doses (MAD) | Placebo Low MAD | DM-101 High MAD | Placebo High MAD | DM-101 2-Day Ultra-Rush Dose Escalation | Placebo 2-Day Ultra-Rush Dose Escalation
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 1/6 | 0/2 | 0/6 | 0/2 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2 | 6/6 | 2/2 | 6/6 | 2/2 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DM-101 Single Dose (N=4) | Placebo Single Dose (N=2) | DM-101 Low Multiple Ascending Doses (MAD) (N=6) | Placebo Low MAD (N=2) | DM-101 High MAD (N=6) | Placebo High MAD (N=2) | DM-101 2-Day Ultra-Rush Dose Escalation (N=4) | Placebo 2-Day Ultra-Rush Dose Escalation (N=1)
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DM-101 Single Dose (N=4) | Placebo Single Dose (N=2) | DM-101 Low Multiple Ascending Doses (MAD) (N=6) | Placebo Low MAD (N=2) | DM-101 High MAD (N=6) | Placebo High MAD (N=2) | DM-101 2-Day Ultra-Rush Dose Escalation (N=4) | Placebo 2-Day Ultra-Rush Dose Escalation (N=1)
Leucocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjuctival Hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Nictitating Spasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 4 (4) | 0 (0) | 6 (6) | 0 (0) | 6 (6) | 0 (0) | 4 (4) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 6 (6) | 0 (0) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling Face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter Site Pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Forced Respiratory Volume Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Hyperreflexia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Orypharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT04266028/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT04266028/SAP_001.pdf